CLINICAL TRIAL: NCT04823416
Title: Risk Factors for Mortality in Cases of Obstructed Left Colonic Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.19.04.169.R1-2019/06/27
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Risk Factors for Mortality in Cases of Obstructed Left Colonic Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stoma (Active Comparator)
  Interventions: Procedure: Stoma
- Resection and stoma (Active Comparator)
  Interventions: Procedure: Resection; Procedure: Stoma

INTERVENTIONS:
Procedure: Resection — Left hemicolectomy
  Arms: Resection and stoma
Procedure: Stoma — Colostomy

SUMMARY:
seeking to identify risk factors leading to mortality in obstructed left cancer colon

ELIGIBILITY:
Inclusion Criteria:

* Patient aged above 18 years admitted at Mansoura University Hospitals complaining from intestinal obstruction due to obstructed left sided carcinoma.

Exclusion Criteria:

* Treatment with non-surgical intervention or spontaneous relief of obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Risk Factors for Mortality in cases of obstructed left colonic Carcinoma | 30 days after surgery
  Predictors of mortality after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Eldakahlia, Egypt